CLINICAL TRIAL: NCT02974491
Title: Acute Consumption of Fuji Apple Juice Does Not Affect Oxidative Stress Biomarkers in Hemodialysis Patients: A Pilot Intervention Study
Brief Title: Consumption of Apple Juice in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Santa Catarina (Other)
Responsible Party: Principal Investigator, Andréia G. Giaretta, principal investigator, Universidade Federal de Santa Catarina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 37090614.6.0000.0118
Record Dates: First submitted 2016-11-10; First posted 2016-11-28 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Oxidative Stress
Keywords: hemodialysis; diabetes mellitus; apple juice; potassium
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Apple Juice (Experimental)
  Interventions: Other: Fuji apple juice

INTERVENTIONS:
Other: Fuji apple juice — On two different days, each volunteer consumed 300 mL Fuji apple juice (AJ), immediately after a dialysis section. After a washout period of 3 weeks, the volunteers drank 150 mL Fuji AJ in a similar manner as described above. Before and after 30 and 60 min of AJ consumption, blood samples were withdrawn for biochemical analysis.

SUMMARY:
The investigators hypothesized that acute consumption of Fuji apple juice (AJ) could increase the antioxidant status and/or decrease the oxidative stress (OS) biomarkers, without increasing serum biochemical parameters in patients undergoing maintenance hemodialysis (MHD). In this pre-post pilot feasibility study, patients served as their own controls, received 300 and 150 mL AJ immediately after a dialysis section, on different days, with a 3 week-washout period. Blood was collected at the baseline period, after 30 and 60 min of AJ consumption. OS biomarkers (total antioxidant status (TAS), total oxidant status (TOS), ascorbic acid, catalase (CAT), glutathione peroxidase (Gpx), superoxide dismutase (SOD) and reduced glutathione (GSH) and potassium, phosphorus, uric acid, and glucose concentrations were analyzed.

DETAILED DESCRIPTION:
Subjects and study design

In this pre-post pilot feasibility study, subjects served as their own controls. Participants were recruited from a hemodialysis clinic, located in Florianópolis' metropolitan area, Santa Catarina state (Southern Brazil), from June to August 2015 with the following inclusion criteria: hemodialysis treatment ≥ 3 months, age ≥ 20 years, and body mass index (BMI) ≥ 23 kg/m2. Exclusion criteria were allergy to apple, presence of cancer or acquired immunodeficiency syndrome, kidney transplant less than 6 months before enrolling in the study, taking antioxidant or nutritional supplements during the 30 days before enrollment, having been hospitalized within 6 weeks before the beginning of the study, or suffering from an acute illness.

Subjects were instructed to keep their usual dietary habits for the duration of the study, except for avoiding intake of polyphenol-rich foods (i.e., vegetables, fruits and fruit-containing products, chocolate, tea, coffee, honey, and any alcoholic beverage) within 2 days before and during intervention. On two different days, each volunteer consumed 300 mL Fuji AJ, immediately after a dialysis section. After a washout period of 3 weeks, the volunteers drank 150 mL Fuji AJ in a similar manner as described above. Before and after 30 and 60 min of AJ consumption, blood samples were withdrawn for biochemical analysis. This protocol was chosen taking into account the previous favorable effects of AJ consumption on serum OS biomarkers described for healthy volunteers.

Baseline clinical and biochemical data were obtained from medical records. This study was approved by the ethics committee of human research of the Federal University of Santa Catarina (UFSC) (protocol number 37090614.6.0000.0118) and all participants gave written and informed consent.

Apple juice and analysis

Fuji apples were obtained from the Experimental Seasonal Fields at the Empresa de Pesquisa Agropecuária e Extensão Rural de Santa Catarina' Station in the city of São Joaquin, Santa Catarina, Brazil (latitude 28º 17' 39", longitude 49º 55' 56" and altitude 1.415 m), harvested in their commercial maturation stage during 2015's harvest. After harvest, apples were stored at 4 ± 1°C. To allow for a quick and easy apple intake in large amounts, 300 mL of AJ, equivalent to 3.5 apples, and 150 mL AJ, equivalent to 1.5 apples were used. Before preparing the juice, the fruits were sanitized in sodium hypochlorite. Apples with peel and no seeds were blended in a centrifugal juice extractor without water addition. Each dose of AJ was prepared and consumed immediately.

The contents of dry matter, total soluble solids, potential of hydrogen (pH) and titratable acidity of AJ were measured following official methods. The total phenolic content of the AJ extracts was measured using the Folin-Ciocalteu method colorimetric. The total flavanol content was estimated using p-dimethylaminocinnamaldehyde (DMACA) method. The total antioxidant capacity was determined using the DPPH (2,2-diphenyl-1-picryl-hydrazyl-hydrate) method. For total monomeric anthocyanin, a spectrophotometric pH differential method was used. Analyses were conducted with each AJ used in the two intervention days, in triplicate.

Blood sampling and laboratory methods

In each experiment day, blood samples from participants were collected in three different moments. Venous blood samples were collected using a vacuum system (Vacutainer Becton Dickinson BD®, São Paulo, Brazil) into heparin, Ethylenediaminetetraacetic acid (EDTA)-containing tubes or additive-free tubes. Plasma and serum were immediately obtained by centrifugation (3,000 revolutions per minute (RPM), 10 min, room temperature) for the measurement of uric acid, phosphorus, glucose, potassium, Total Antioxidant Status (TAS) and Total Oxidant Status( TOS). In order to quantify the endogenous antioxidant enzymes, an aliquot of whole blood was lysed. In order to measure reduced glutathione (GSH), an aliquot of whole blood was preserved in N-ethylmaleimide (NEM). All samples were immediately stored at -80°C for later analysis in duplicate.

Serum uric acid, phosphorus and glucose concentrations were determined using commercially available kits (Labtest Diagnóstica SA, Lagoa Santa, Minas Gerais, Brazil) in an automated multi-biochemical analyzer (Cobas Miras Plus, Roche®, Germany). Serum potassium levels were measured in an automated Dimension Max System (Siemens Healthcare Diagnostics Products®, Germany), according to the manufacturer's instructions.

TAS and TOS assays were measured spectrophotometrically, according to Erel's methods. Ascorbic acid and GSH were determined using high-performance liquid chromatography (HPLC), as previously described. The superoxide dismutase (SOD) activity was evaluated using SOD Assay Kit (Sigma Aldrich®, St. Louis, Missouri, USA) according to the manufacturer's instructions. Catalase (CAT) activity was determined spectrophotometrically according to the previously described method. The glutathione peroxidase (GPx) activity was determined using the NADPH oxidation rate method.

ELIGIBILITY:
Inclusion Criteria:

* hemodialysis treatment ≥ 3 months, age ≥ 20 years, and body mass index ≥ 23 kg/m2

Exclusion Criteria:

* allergy to apple, presence of cancer or acquired immunodeficiency syndrome, kidney transplant less than 6 months before enrolling in the study, taking antioxidant or nutritional supplements during the 30 days before enrollment, having been hospitalized within 6 weeks before the beginning of the study, or suffering from an acute illness

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Measuring oxidative stress biomarkers | Change from baseline at 30 and 60 minutes
  Total antioxidant status (TAS) (mmol/L) and total oxidant status (TOS) (mmol/L) was measured at the baseline period, after 30 and 60 min of acute consumption of 300 and 150 mL of Fuji apple (Malus domestica Borkh) juice. Patients were not fasted for the withdrawal of blood. This measure was taken to prevent discomfort among volunteers. Venous blood samples were collected through aseptic venipuncture on the opposite arm of the arteriovenous fistula by a qualified professional using a vacuum system into heparin or EDTA-containing tubes or tubes without additives according to established standards of clinical and biological safety.
Measuring endogenous antioxidant enzymes | Change from baseline at 30 and 60 minutes
  Catalase (U mg/Hb), glutathione peroxidase (U mg/Hb) and superoxide dismutase (U mg/Hb) was measured at the baseline period, after 30 and 60 min of acute consumption of 300 and 150 mL of Fuji apple (Malus domestica Borkh) juice. Patients were not fasted for the withdrawal of blood. This measure was taken to prevent discomfort among volunteers. Venous blood samples were collected through aseptic venipuncture on the opposite arm of the arteriovenous fistula by a qualified professional using a vacuum system into heparin or EDTA-containing tubes or tubes without additives according to established standards of clinical and biological safety.
Measuring oxidative stress biomarkers | Change from baseline at 30 and 60 minutes
  Ascorbic acid (micromole/L) was measured at the baseline period, after 30 and 60 min of acute consumption of 300 and 150 mL of Fuji apple (Malus domestica Borkh) juice. Patients were not fasted for the withdrawal of blood. This measure was taken to prevent discomfort among volunteers. Venous blood samples were collected through aseptic venipuncture on the opposite arm of the arteriovenous fistula by a qualified professional using a vacuum system into heparin or EDTA-containing tubes or tubes without additives according to established standards of clinical and biological safety.
Measuring oxidative stress biomarkers | Change from baseline at 30 and 60 minutes
  Reduced glutathione (micromole mg/Hb) was measured at the baseline period, after 30 and 60 min of acute consumption of 300 and 150 mL of Fuji apple (Malus domestica Borkh) juice. Patients were not fasted for the withdrawal of blood. This measure was taken to prevent discomfort among volunteers. Venous blood samples were collected through aseptic venipuncture on the opposite arm of the arteriovenous fistula by a qualified professional using a vacuum system into heparin or EDTA-containing tubes or tubes without additives according to established standards of clinical and biological safety.
Measuring serum biochemical parameters | Change from baseline at 30 and 60 minutes
  Potassium (mmol/L), phosphorus (mmol/L) and glucose (mmol/L) was measured at the baseline period, after 30 and 60 min of acute consumption of 300 and 150 mL of Fuji apple (Malus domestica Borkh) juice. Patients were not fasted for the withdrawal of blood. This measure was taken to prevent discomfort among volunteers. Venous blood samples were collected through aseptic venipuncture on the opposite arm of the arteriovenous fistula by a qualified professional using a vacuum system into heparin or EDTA-containing tubes or tubes without additives according to established standards of clinical and biological safety.
Measuring serum biochemical parameters | Change from baseline at 30 and 60 minutes
  Uric acid (micromole/L) was measured at the baseline period, after 30 and 60 min of acute consumption of 300 and 150 mL of Fuji apple (Malus domestica Borkh) juice. Patients were not fasted for the withdrawal of blood. This measure was taken to prevent discomfort among volunteers. Venous blood samples were collected through aseptic venipuncture on the opposite arm of the arteriovenous fistula by a qualified professional using a vacuum system into heparin or EDTA-containing tubes or tubes without additives according to established standards of clinical and biological safety.
Evaluating heigth | at baseline
  Height (meters) data were obtained from the patient's files.
Evaluating weight | At baseline
  Weight (kilograms) data were obtained from the patient's files.
Evaluating body mass index | At baseline
  Body mass index (BMI) (Kg/m2) data were obtained from the patient's files.
Evaluating medication | At baseline
  Medication data were obtained from the patient's files.
Evaluating adequacy of the dialysis treatment | At baseline
  Adequacy of the dialysis treatment was captured by extracting the routine Kt/V from the medical record.

REFERENCES:
- [Background] Ruskovska T, Jansen EH, Antarorov R. Evaluation of assays for measurement of serum (anti)oxidants in hemodialysis patients. Biomed Res Int. 2014;2014:843157. doi: 10.1155/2014/843157. Epub 2014 May 19. PMID 24982909
- [Background] Halliwell, B, Gutteridge, JMC. Cellular responses to oxidative stress: adaptation, damage, repair, senescence and death. In: Halliwell, B, Gutteridge, JMC. Free Radical in Biology and Medicine. 4th ed. Oxford, UK: Oxford University Press; 2007, p. 87-267.
- [Background] McDonald CI, Fraser JF, Coombes JS, Fung YL. Oxidative stress during extracorporeal circulation. Eur J Cardiothorac Surg. 2014 Dec;46(6):937-43. doi: 10.1093/ejcts/ezt637. Epub 2014 Jan 30. PMID 24482384
- [Background] Melidou M, Riganakos K, Galaris D. Protection against nuclear DNA damage offered by flavonoids in cells exposed to hydrogen peroxide: the role of iron chelation. Free Radic Biol Med. 2005 Dec 15;39(12):1591-600. doi: 10.1016/j.freeradbiomed.2005.08.009. Epub 2005 Aug 29. PMID 16298684
- [Background] Spormann TM, Albert FW, Rath T, Dietrich H, Will F, Stockis JP, Eisenbrand G, Janzowski C. Anthocyanin/polyphenolic-rich fruit juice reduces oxidative cell damage in an intervention study with patients on hemodialysis. Cancer Epidemiol Biomarkers Prev. 2008 Dec;17(12):3372-80. doi: 10.1158/1055-9965.EPI-08-0364. PMID 19064553
- [Background] Castilla P, Echarri R, Davalos A, Cerrato F, Ortega H, Teruel JL, Lucas MF, Gomez-Coronado D, Ortuno J, Lasuncion MA. Concentrated red grape juice exerts antioxidant, hypolipidemic, and antiinflammatory effects in both hemodialysis patients and healthy subjects. Am J Clin Nutr. 2006 Jul;84(1):252-62. doi: 10.1093/ajcn/84.1.252. PMID 16825703
- [Background] Shema-Didi L, Sela S, Ore L, Shapiro G, Geron R, Moshe G, Kristal B. One year of pomegranate juice intake decreases oxidative stress, inflammation, and incidence of infections in hemodialysis patients: a randomized placebo-controlled trial. Free Radic Biol Med. 2012 Jul 15;53(2):297-304. doi: 10.1016/j.freeradbiomed.2012.05.013. Epub 2012 May 17. PMID 22609423
- [Background] Fouque D, Kalantar-Zadeh K, Kopple J, Cano N, Chauveau P, Cuppari L, Franch H, Guarnieri G, Ikizler TA, Kaysen G, Lindholm B, Massy Z, Mitch W, Pineda E, Stenvinkel P, Trevino-Becerra A, Wanner C. A proposed nomenclature and diagnostic criteria for protein-energy wasting in acute and chronic kidney disease. Kidney Int. 2008 Feb;73(4):391-8. doi: 10.1038/sj.ki.5002585. Epub 2007 Dec 19. PMID 18094682
- [Background] Golding JB, McGlasson WB, Wyllie SG, Leach DN. Fate of apple peel phenolics during cool storage. J Agric Food Chem. 2001 May;49(5):2283-9. doi: 10.1021/jf0015266. PMID 11368590
- [Background] Dai X, Luo H, Jiang L, Ling L, Xue Y, Yu Z. Efficacy of different sanitizing agents and their combination on microbe population and quality of fresh-cut Chinese chives. J Food Sci. 2012 Jul;77(7):M348-53. doi: 10.1111/j.1750-3841.2012.02770.x. Epub 2012 Jun 18. PMID 22708729
- [Background] Association of Official Analytical Chemists (AOAC). Official Methods of Analysis. 18th ed. Washington, DC: Association of Official Analytical Chemists; 2005.
- [Background] Singleton, VL, Rossi, JA. Colorimetry of total phenolics with phosphomolybdic phosphotungstic acid reagents. Am J Enol Vitic 1965;16(3):144-58.
- [Background] Arnous, A, Markis, D, Kefalas, P. Correlation of pigment and flavonol content with antioxidant properties in selected aged regional wines from Greece. J Food Composit Ana 2002;15(6):655-65.
- [Background] Brand-Williams, W, Cuvelier, ME, Berset, C. Use of free radical method to evaluate antioxidant activity. LWT Food Sci Technol 1995;28(1):25-30.
- [Background] Giusti, MM, Wrolstad, RE. Anthocyanins: characterization and measurement with UV-visible spectroscopy. In: Wrolstald, RE, ed. Current Protocols in Food Analytical Chemistry. New York, NY: John Wiley and Sons; 2001, p. 1-13.
- [Background] Erel O. A novel automated direct measurement method for total antioxidant capacity using a new generation, more stable ABTS radical cation. Clin Biochem. 2004 Apr;37(4):277-85. doi: 10.1016/j.clinbiochem.2003.11.015. PMID 15003729
- [Background] Erel O. A new automated colorimetric method for measuring total oxidant status. Clin Biochem. 2005 Dec;38(12):1103-11. doi: 10.1016/j.clinbiochem.2005.08.008. Epub 2005 Oct 7. PMID 16214125
- [Background] Chung WY, Chung JK, Szeto YT, Tomlinson B, Benzie IF. Plasma ascorbic acid: measurement, stability and clinical utility revisited. Clin Biochem. 2001 Nov;34(8):623-7. doi: 10.1016/s0009-9120(01)00270-3. PMID 11849621
- [Background] Giustarini D, Dalle-Donne I, Milzani A, Fanti P, Rossi R. Analysis of GSH and GSSG after derivatization with N-ethylmaleimide. Nat Protoc. 2013 Sep;8(9):1660-9. doi: 10.1038/nprot.2013.095. Epub 2013 Aug 1. PMID 23928499
- [Background] Johansson LH, Borg LA. A spectrophotometric method for determination of catalase activity in small tissue samples. Anal Biochem. 1988 Oct;174(1):331-6. doi: 10.1016/0003-2697(88)90554-4. PMID 3064653
- [Background] Wendel A. Glutathione peroxidase. Methods Enzymol. 1981;77:325-33. doi: 10.1016/s0076-6879(81)77046-0. No abstract available. PMID 7329310
- [Background] National Kidney Foundation. K/DOQI clinical practice guidelines for bone metabolism and disease in chronic kidney disease. Am J Kidney Dis. 2003 Oct;42(4 Suppl 3):S1-201. No abstract available. PMID 14520607
- [Background] Ceriello A, Colagiuri S. International Diabetes Federation guideline for management of postmeal glucose: a review of recommendations. Diabet Med. 2008 Oct;25(10):1151-6. doi: 10.1111/j.1464-5491.2008.02565.x. PMID 19046192